CLINICAL TRIAL: NCT00743171
Title: Long-Term Study On Home Spirometry After Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Jens Gottlieb, Hannover Medical School, Dpt. Pneumology
Other Study IDs: MHH 2008-3
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Lung Transplantation; Rejection; Death; Bronchiolitis Obliterans
Keywords: Lung transplantation; Home spirometry; non-adherence; outcomes; bronchiolitis obliterans
MeSH Terms: conditions — Rejection, Psychology; Death; Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Good adherent patient: patient performed ≥ 80% of predicted HS within 24 months
- 2: Moderate adherent patient: patient performed ≥ 50% of predicted HS within 24 months
- 3: Non-adherent patient: patient performed < 50% of predicted HS within 24 months.

SUMMARY:
Prospective cohort, mono-center study included electronic data of home spirometry (HS, lung function) of lung transplant recipients

DETAILED DESCRIPTION:
Study period between 1/2/2000 and 31/12/2003 Follow-up until 31/12/2007

Patient will be stratified according to adherence to HS during the first 2 postoperative years Good adherent patient: patient performed ≥ 80% of predicted HS within 24 months Moderate adherent patient: patient performed ≥ 50% of predicted HS within 24 months Non-adherent patient: patient performed < 50% of predicted HS within 24 months.

Primary outcome measure graft loss at end of follow-up

Secondary outcome measure number of acute rejections during follow-up number of hospitalisation during follow-up Incidence of bronchiolitis obliterans syndrome during follow-up

ELIGIBILITY:
Inclusion Criteria:

* Any type of lung transplant incl single, double, combined and re-do
* > 18 years of age
* LTx or HLTx ≥ 6mts post Tx
* Stable health condition at study entry (pt stays within home environment)
* Sufficient language skills for AMOS training
* Successful AMOS training
* Follow-up at our center (≥6 mts post LTx)
* Willingness to participate by informed consent

Exclusion Criteria:

* Refused consent
* BOS diagnosis before study inclusion
* Malignancy before study inclusion
* Loss for follow-up (≤ 6 mts after study inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung transplant recipients surviving to outpatient follow-up >6 months in Hannover Medical School
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2000-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Graft loss | 3 year

SECONDARY OUTCOMES:
BOS | 3 year
Number of acute rejections | 3 year
Number of hospitalizations | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Jens T Gottlieb, MD, Principal Investigator — Dpt. Pneumology; Christiane Kugler, MSc, Principal Investigator — Dpt. Cardiothoracic, Transplantation and Vascular Surgery
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Background] Finkelstein SM, Scudiero A, Lindgren B, Snyder M, Hertz MI. Decision support for the triage of lung transplant recipients on the basis of home-monitoring spirometry and symptom reporting. Heart Lung. 2005 May-Jun;34(3):201-8. doi: 10.1016/j.hrtlng.2004.09.003. PMID 16015225
- [Background] Dew MA, Dimartini AF, De Vito Dabbs A, Zomak R, De Geest S, Dobbels F, Myaskovsky L, Switzer GE, Unruh M, Steel JL, Kormos RL, McCurry KR. Adherence to the medical regimen during the first two years after lung transplantation. Transplantation. 2008 Jan 27;85(2):193-202. doi: 10.1097/TP.0b013e318160135f. PMID 18212623
- [Background] De Geest S, Dobbels F, Fluri C, Paris W, Troosters T. Adherence to the therapeutic regimen in heart, lung, and heart-lung transplant recipients. J Cardiovasc Nurs. 2005 Sep-Oct;20(5 Suppl):S88-98. doi: 10.1097/00005082-200509001-00010. PMID 16160588
- [Background] Finkelstein SM, Snyder M, Edin-Stibbe C, Chlan L, Prasad B, Dutta P, Lindgren B, Wielinski C, Hertz MI. Monitoring progress after lung transplantation from home-patient adherence. J Med Eng Technol. 1996 Nov-Dec;20(6):203-10. doi: 10.3109/03091909609008999. PMID 9029392
- [Background] Bjortuft O, Johansen B, Boe J, Foerster A, Holter E, Geiran O. Daily home spirometry facilitates early detection of rejection in single lung transplant recipients with emphysema. Eur Respir J. 1993 May;6(5):705-8. PMID 8390943